CLINICAL TRIAL: NCT03577171
Title: A Phase 2a, Multi-center, Double-blind, Placebo-controlled Study Evaluating ABI-H0731+ Entecavir vs Entecavir Alone for the Treatment of Viremic HBeAg-positive Patients With Chronic Hepatitis B
Brief Title: A Study Evaluating ABI-H0731+ Entecavir vs Entecavir Alone for the Treatment of Viremic HBeAg-positive Participants With Chronic Hepatitis B Virus Infection (cHBV)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assembly Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ABI-H0731-202
Record Dates: First submitted 2018-06-06; First posted 2018-07-05 (Actual); Results first posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Chronic Hepatitis B
Keywords: cHBV; HBV; HBeAg-positive; hepatitis B; vebicorvir; VBR
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — entecavir

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ABI-H0731 + SOC ETV (Experimental): Participants with cHBV who are currently not being treated will receive ABI-H0731 along with SOC ETV tablets orally for 24 weeks. Eligible participants may enter a separate extension study after Week 24 to continue open-label ABI-H0731 for up to an additional year if necessary.
  Interventions: Drug: ABI-H0731; Drug: SOC ETV
- Placebo + SOC ETV (Experimental): Participants with cHBV who are currently not being treated will receive matching placebo along with SOC ETV tablets orally for 24 weeks. Eligible participants may enter a separate extension study after Week 24 to start treatment on open-label ABI-H0731 for up to a year if necessary.
  Interventions: Drug: SOC ETV; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: ABI-H0731 — Participants will receive 300mg QD of ABI-H0731 tablets orally.
  Arms: ABI-H0731 + SOC ETV
Drug: SOC ETV — Participants will receive SOC ETV (0.5 mg QD) orally as per approved package insert.
  Other Names: Entecavir
Drug: Placebo Oral Tablet — Participants will receive matching QD placebo tablets orally.
  Arms: Placebo + SOC ETV

SUMMARY:
The purpose of this study is to determine if ABI-H0731 given in combination with a standard of care (SOC) entecavir (ETV) is safe and effective in participants with chronic hepatitis B infection (cHBV)

DETAILED DESCRIPTION:
This is a Phase 2a, multi-center, double-blind, placebo-controlled study evaluating ABI-H0731+ ETV vs ETV alone for the treatment of viremic hepatitis B "e" antigen (HBeAg)-positive participants with cHBV.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female between ages 18 and 70 years
* HBeAg-positive at screening
* In good general health except for cHBV
* HBV viral load ≥2×105 IU/mL
* Hepatitis B surface antigen (HBsAg) >1000 IU/mL at screening

Key Exclusion Criteria:

* Any prior treatment with lamivudine or telbivudine, previous treatment with an investigational agent for HBV other than ABI-H0731; or any other SOC treatment for >4 weeks
* Co-infection with HIV, hepatitis C virus (HCV), hepatitis E virus (HEV) or hepatitis D virus (HDV)
* History or evidence of hepatic decompensation (including gastrointestinal bleeding or esophageal varices) at any time prior to or at time of screening
* Clinically significant cardiac or pulmonary disease, chronic or recurrent renal or urinary tract disease, liver disease other than HBV, endocrine disorder, autoimmune disorder, diabetes mellitus requiring treatment with insulin or hypoglycemic agents, neuromuscular, musculoskeletal, or mucocutaneous conditions requiring frequent treatment, seizure disorders requiring treatment, or other medical conditions requiring frequent medical management or pharmacologic or surgical treatment that in the opinion of the Investigator or the Sponsor makes the participant unsuitable for the study
* Previous treatment with an investigational agent for HBV other than ABI-H0731 in the last 6 months before screening
* History of hepatocellular carcinoma (HCC)
* Females who are lactating or pregnant or wish to become pregnant are excluded from the study
* Exclusionary laboratory parameters at screening:

  * Platelet count <100,000/mm3
  * Albumin <lower limit of normal (LLN)
  * Direct bilirubin >1.2×upper limit of normal (ULN)
  * Alanine aminotransferase (ALT) >10×ULN at screening
  * Serum alpha fetoprotein (AFP) ≥100 ng/mL. If AFP at Screening is >ULN but <100 ng/mL, participant is eligible if a hepatic imaging study prior to the initiation of study drug reveals no lesions suspicious of possible HCC
  * International Normalized Ratio (INR) >1.5×ULN
  * Glomerular filtration rate (GFR) <60 mL/min/1.73 m2 by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (7):
  - Southern California Research Center, Coronado, California
  - Asia Pacific Liver Center, Los Angeles, California
  - Research and Education, San Diego, California
  - Quest Clinical Research, San Francisco, California
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - NYU Langone Health, New York, New York
  - Xiaoli Ma MD, Philadelphia, Pennsylvania
- Canada (2):
  - GI Research Institute, Vancouver, British Columbia
  - Toronto Liver Center, Toronto, Ontario
- University of Hong Kong, Queen Mary Hospital, Hong Kong, Hong Kong
- Waikato Hospital, Hamilton, New Zealand
- King's College London, London, United Kingdom

REFERENCES:
- [Derived] Sulkowski MS, Agarwal K, Ma X, Nguyen TT, Schiff ER, Hann HL, Dieterich DT, Nahass RG, Park JS, Chan S, Han SB, Gane EJ, Bennett M, Alves K, Evanchik M, Yan R, Huang Q, Lopatin U, Colonno R, Ma J, Knox SJ, Stamm LM, Bonacini M, Jacobson IM, Ayoub WS, Weilert F, Ravendhran N, Ramji A, Kwo PY, Elkhashab M, Hassanein T, Bae HS, Lalezari JP, Fung SK, Yuen MF. Safety and efficacy of vebicorvir administered with entecavir in treatment-naive patients with chronic hepatitis B virus infection. J Hepatol. 2022 Nov;77(5):1265-1275. doi: 10.1016/j.jhep.2022.05.027. Epub 2022 Jun 11. PMID 35697332

RESULTS

PARTICIPANT FLOW:
Groups:
- ABI-H0731 + SOC ETV: Participants with chronic hepatitis B infection (cHBV) who are currently not being treated will receive ABI-H0731 along with standard of care (SOC) entecavir (ETV) tablets orally for 24 weeks. Eligible participants may enter a separate extension study after Week 24 to continue open-label ABI-H0731 for up to an additional year if necessary.
  ABI-H0731: Participants will receive 300mg QD of ABI-H0731 tablets orally.
  SOC ETV: Participants will receive SOC ETV (0.5 mg QD) orally as per approved package insert.
Period: Overall Study
Arm/Group | ABI-H0731 + SOC ETV | Placebo + SOC ETV
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | ABI-H0731 + SOC ETV | Placebo + SOC ETV | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (14.13) | 34.1 (11.39) | 34.9 (12.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 12 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 11 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  New Zealand | 1 | 0 | 1
  Canada | 1 | 2 | 3
  Hong Kong | 3 | 2 | 5
  United States | 7 | 7 | 14
  United Kingdom | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean log10 HBV DNA From Baseline (Day 1) to Week 12 or Week 24 on ABI H0731 + SOC ETV as Compared to Placebo + SOC ETV
Description: Hepatitis B virus (HBV) DNA was measured using COBAS TaqMan Version 2.0. The lower limit of quantitation (LLOQ) was 20 IU/mL and the limit of detection (LOD) was 10 IU/mL.
Time Frame: Baseline, Week 12, and Week 24
Population: Intent-to-treat (ITT) population: all randomized participants
Measure: Mean (Standard Deviation); unit: Log10 International Units (IU)/mL
Arm/Group | ABI-H0731 + SOC ETV | Placebo + SOC ETV
Number analyzed (Participants) | 13 | 12
Log10 International Units (IU)/mL
  Baseline | 7.91 (0.890) | 8.03 (0.999)
  Change from Baseline at Week 12 | -4.45 (1.027) | -3.30 (1.182)
  Change from Baseline at Week 24 | -5.33 (1.594) | -4.20 (0.976)
Statistical Analysis 1: Comparison: ABI-H0731 + SOC ETV vs Placebo + SOC ETV; Least Squares (LS) Mean Difference ABI-H0731 + SOC ETV minus Placebo + SOC ETV at Week 12; Test type: Other; p = 0.0077, Repeated measures analysis; LS Mean Difference = -1.154, 95% CI 2-sided [-1.986 to -0.322]
Statistical Analysis 2: Comparison: ABI-H0731 + SOC ETV vs Placebo + SOC ETV; Least Squares Mean Difference ABI-H0731 + SOC ETV minus Placebo + SOC ETV at Week 24; Test type: Other; p = 0.0084, Repeated measures analysis; LS Mean Difference = -1.141, 95% CI 2-sided [-1.973 to -0.309]

2. Secondary Outcome: Number of Participants One or More Adverse Events
Time Frame: Up to Follow-up (maximum up to Week 36)
Population: Safety population: all randomized participants who received any amount of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | ABI-H0731 + SOC ETV | Placebo + SOC ETV
Number analyzed (Participants) | 13 | 12
Participants | 7 | 5

3. Secondary Outcome: Number of Participants With Premature Study Discontinuation
Time Frame: Up to Follow-up (maximum up to Week 36)
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | ABI-H0731 + SOC ETV | Placebo + SOC ETV
Number analyzed (Participants) | 13 | 12
Participants | 0 | 0

4. Secondary Outcome: Number of Participants With One or More Abnormal Safety Laboratory Result
Time Frame: Up to Week 36
Population: Safety population: all randomized participants who received any amount of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | ABI-H0731 + SOC ETV | Placebo + SOC ETV
Number analyzed (Participants) | 13 | 12
Participants | 8 | 10

5. Secondary Outcome: Number of Participants With a Clinically-significant Electrocardiogram Abnormality
Time Frame: Up to Week 24
Population: Safety population: all randomized participants who received any amount of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | ABI-H0731 + SOC ETV | Placebo + SOC ETV
Number analyzed (Participants) | 13 | 12
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With a Clinically-significant Change in Vital Signs
Description: Vital signs assessed were body temperature, respiratory rate, and pulse rate
Time Frame: Baseline and up to Week 24
Population: Safety population: all randomized participants who received any amount of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | ABI-H0731 + SOC ETV | Placebo + SOC ETV
Number analyzed (Participants) | 13 | 12
Participants | 0 | 0

7. Secondary Outcome: Number of Participants With Abnormal Alanine Aminotransferase (ALT) at Baseline Who Have Normal ALT at Week 24 on ABI-H0731 + SOC ETV as Compared to Placebo + SOC ETV
Time Frame: Baseline to Week 24
Population: Participants in the ITT population with abnormal ALT at Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | ABI-H0731 + SOC ETV | Placebo + SOC ETV
Number analyzed (Participants) | 4 | 4
Participants | 4 | 2

8. Secondary Outcome: Number of Participants With a Decline in Viral DNA to Below Limit of Quantitation on ABI-H0731 + SOC ETV as Compared to Placebo + SOC ETV
Description: HBV DNA was measured using COBAS TaqMan Version 2.0. The LLOQ was 20 IU/mL and the LOD was 10 IU/mL. The number of participants with HBV DNA below the limit of quantitation (<20 IU/mL) and target detected (≥10 IU/mL) was assessed.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, and 24
Population: ITT population and had viral DNA data available
Measure: Count of Participants; unit: Participants
Arm/Group | ABI-H0731 + SOC ETV | Placebo + SOC ETV
Number analyzed (Participants) | 13 | 12
Participants
  Baseline | 0 | 0
  Week 2 | 0 | 0
  Week 4 | 0 | 0
  Week 8 | 1 | 0
  Week 12 | 1 | 0
  Week 16: number analyzed (Participants) | 11 | 11
  Week 16 | 2 | 0
  Week 20 | 1 | 1
  Week 24 | 3 | 1

9. Secondary Outcome: Median Time to Viral Suppression, Defined as HBV DNA <20 IU/mL, on ABI-H0731 + ETV as Compared to Placebo + ETV
Description: Median time to viral suppression will be calculated and evaluated between participants on ABI-H0731 + ETV as compared to placebo + ETV.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, and 24
Population: Median time to viral suppression could not be calculated because fewer than 50% of participants achieved viral suppression within 24 weeks.
Arm/Group | ABI-H0731 + SOC ETV | Placebo + SOC ETV
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Number of Participants With Emergence of Resistant HBV Variants on ABI-H0731 + SOC ETV as Compared to Placebo + SOC ETV
Description: Emergence of a resistant HBV variant was defined as an increase of ≥1 log10 IU/mL from the nadir in HBV DNA.
Time Frame: Up to Week 36
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | ABI-H0731 + SOC ETV | Placebo + SOC ETV
Number analyzed (Participants) | 13 | 12
Participants
  Emergence of resistant HBV variants | 1 | 1
  No emergence of resistant HBV variants | 12 | 11

11. Secondary Outcome: Trough Levels of ABI-H0731 on ABI-H0731 + SOC ETV Therapy
Time Frame: Before dosing at Baseline (Day 1), Weeks 2, 4, 12, and 24
Population: Results were analyzed and reported only for participants in the safety population who received ABI-H0731 + SOC ETV and had ABI-H0731 pharmacokinetic data assessments available.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ABI-H0731 + SOC ETV
Number analyzed (Participants) | 13
ng/mL
  Baseline (Day 1) | NA (NA) — Plasma levels for all participants were below the limit of quantitation
  Week 2 | 1480 (458)
  Week 4 | 1290 (434)
  Week 12 | 1270 (413)
  Week 24 | 1470 (547)

12. Secondary Outcome: Trough Levels of ETV on ABI-H0731 + ETV Therapy as Compared With Placebo + ETV Therapy
Time Frame: Before dosing at Baseline (Day 1), Weeks 2, 4, 12, and 24
Population: Results were analyzed and reported only for participants in the safety population who had ETV pharmacokinetic data assessments available.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ABI-H0731 + SOC ETV | Placebo + SOC ETV
Number analyzed (Participants) | 13 | 12
ng/mL
  Baseline (Day 1): number analyzed (Participants) | 12 | 12
  Baseline (Day 1) | 0.00325 (0.0113) | 0 (0)
  Week 2 | 0.432 (0.126) | 0.497 (0.473)
  Week 4: number analyzed (Participants) | 13 | 11
  Week 4 | 0.419 (0.119) | 0.618 (0.736)
  Week 12: number analyzed (Participants) | 12 | 11
  Week 12 | 0.378 (0.149) | 0.666 (0.766)
  Week 24 | 0.411 (0.143) | 0.408 (0.131)

13. Secondary Outcome: Trough to Peak Ratios of ABI-H0731 on ABI-H0731 + ETV Therapy
Time Frame: Baseline, Weeks 2, 4, 12, and 24
Population: Trough to peak ratios were not calculated due to an insufficient number of optional peak exposure samples.
Arm/Group | ABI-H0731 + SOC ETV
Number analyzed (Participants) | 0

14. Secondary Outcome: Trough to Peak Ratios of ETV on ABI-H0731 + ETV Therapy as Compared With Placebo + ETV Therapy
Time Frame: Baseline, Weeks 2, 4, 12, 24, and 28
Population: Trough to peak ratios were not calculated due to an insufficient number of optional peak exposure samples.
Arm/Group | ABI-H0731 + SOC ETV | Placebo + SOC ETV
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Week 36
Description: Safety population
Arm/Group | ABI-H0731 + SOC ETV | Placebo + SOC ETV
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 7/13 | 5/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABI-H0731 + SOC ETV (N=13) | Placebo + SOC ETV (N=12)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (2)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2)
Electrocardiogram T wave abnormal (Investigations) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Assembly Biosciences agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Assembly Biosciences supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-06-18): https://cdn.clinicaltrials.gov/large-docs/71/NCT03577171/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/71/NCT03577171/SAP_001.pdf